CLINICAL TRIAL: NCT05776485
Title: Protein Turnover in Healthy and Overuse-diseased Tendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ann Damgaard, Medical Doctor, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Project 159
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Patella; Tendinitis
MeSH Terms: conditions — Patella Fracture; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic tendinopathy patients (Experimental)
  Interventions: Other: Cross-sectional comparison between healthy and tendinopathic group
- Healthy controls (Experimental)
  Interventions: Other: Progressive resistance training; Other: Cross-sectional comparison between healthy and tendinopathic group

INTERVENTIONS:
Other: Progressive resistance training — Only the control group: 3 exercise bouts within the study period. Comparison between exercised and non-exercised leg.
  Arms: Healthy controls
Other: Cross-sectional comparison between healthy and tendinopathic group — Comparison of primary and secondary outcomes.

SUMMARY:
The goal of this clinical trial is to examine the regional protein turnover in tendon tissue from patients with chronic patellar tendinopathy and comparing this to healthy controls. Further we will examine the effect of resistance training on protein turnover in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Physical active men and women
* Body mass index 18,5 - 30 kg/m2

Inclusion Criteria for the chronic tendinopathy group:

* Debut of symptom > 90 days prior to inclusion.
* Subjective activity related pain in patella tendon.
* Clinical symptoms of patella tendinopathy.
* Ultrasound verification of at least 1 in three of the following: Enchanced anterior-posterior diameter, increased Doppler signal and/or a hypoechoic area in the diseased part of the tendon.

Exclusion Criteria for all participants:

* Former knee surgery or injuries to the patella tendon.
* Local injection of corticosteroids within 12 months.
* Medication that affects protein synthesis in tendon tissue.
* Former/current use of anabolic steroids or growth hormone.
* Smoking
* Known rheumatoid disease or diabetes.
* Former participation in trials using deuterated water and 15N tracers.
* Treatment for patella tendinopathy within 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Protein turnover in tendon tissue from patients with chronic tendinopathy compared to healthy controls | 8 days
  Fractional synthesis rate (FSR) measured in % pr. day in the trypsin-soluble and trypsin-insoluble fraction

SECONDARY OUTCOMES:
Tracer incorporation in isolated fractions of the tendon | 8 days
  15N hydroxyproline enrichment measured in Mole percent Excess in the trypsin-soluble and trypsin-insoluble fraction
Tracer incorporation in isolated fractions of the tendon | 8 days
  15N proline enrichment measured in Mole percent Excess in the trypsin-soluble and trypsin-insoluble fraction
Anterior-posterior dimensions of patella tendon | 8 days
  Measured in millimeter
Doppler flow in patella tendon | 8 days
  Classified in grading system from 0-3.
Subjective pain in patella tendon | 8 days
  Questionnaire
Subjective measure of physical activity and function | 1 day
  Questionnaire
Single-leg decline squat test | 1 day
  Subjective pain on a scale from 0-10
One leg knee extension strength test | 8 days
  Only control-group.
Leg press strength test | 8 days
  Only control-group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjær, Professor, Principal Investigator — Institute of Sports Medicine, Copenhagen
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers upon request.